CLINICAL TRIAL: NCT04161157
Title: Piloting Pathways, a Hope-enhancing Intervention to Address Activity and Role Function in Metastatic Lung Cancer Patients
Brief Title: Piloting Pathways With Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laurie McLouth (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Laurie McLouth, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 52168; R03CA235171-01A1 (NIH)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathways (Experimental): Pathways is designed to help patients identify and pursue values-based goals and address potential goal obstacles, including lung cancer stigma.
  Interventions: Behavioral: Pathways

INTERVENTIONS:
Behavioral: Pathways — Goal-setting intervention to help patients identify personal values, value-consistent goals, and ways to pursue goals and address goal obstacles. Although potential refinements may occur based on aim 1 (refining procedures and content with 6 patients), Pathways is designed to consist primarily of 2 in-person sessions (~30-60 minutes) delivered when patients are in clinic for cancer treatment, with supporting phone calls and contact in between sessions.

SUMMARY:
The purpose of this research is to determine the feasibility of a new supportive intervention, called Pathways, for patients with advanced stage and metastatic lung cancer.

DETAILED DESCRIPTION:
In this study, investigators will first test the Pathways procedures with 6 patients to identify any improvements that need to be made. Then, investigators will test the feasibility of the Pathways intervention with 20 patients who are undergoing cancer treatment for advanced stage or metastatic lung cancer. Pathways is designed to help patients set and pursue personal goals during lung cancer treatment. In this study, investigators want to see if they can recruit patients with lung cancer who are being treated at the University of Kentucky Markey Cancer Center to participate in the Pathways intervention.

ELIGIBILITY:
Inclusion Criteria:

* new or recurrent stage IIIB, stage IIIC or stage IV non-small cell lung cancer (NSCLC) or extensive stage SCLC
* 18 years of age or older
* ECOG PS 0-2/Karnofsky 60-100
* 3 to 12 weeks into active cancer treatment

Exclusion Criteria:

* unstable brain metastases
* cognitive or psychiatric condition for which participating would be inappropriate
* unable to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie McLouth, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pathways
Started | 53
Completed | 40
Not Completed | 13
Not completed — Lost to Follow-up | 4
Not completed — Death | 3
Not completed — Ineligible | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: 53 participants were enrolled in the study; however, 1 participant dropped from the study before baseline measures were collected.
Arm/Group | Pathways
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant dropped from the study before baseline measures were collected.
  years | 61.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant dropped from the study before baseline measures were collected.
  Participants
    Female | 31
    Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant dropped from the study before baseline measures were collected.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 52
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 44
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment: Percentage of Eligible and Approached Patients Who Agree to Participate
Description: Percentage of eligible and approached patients who agree to participate
Time Frame: 9 months
Population: 98 potentially eligible people were approached, of whom 53 agreed to participate.
Measure: Count of Participants; unit: Participants
Arm/Group | Pathways
Number analyzed (Participants) | 98
Participants | 53

2. Primary Outcome: Acceptability: Ratings
Description: Mean acceptability ratings on individual items of acceptability developed by study team (e.g., convenience of the intervention, helpfulness of the intervention, relevance of the intervention; scores of at least 7/10 on each item, possible range = 1-10, higher scores indicate higher acceptability).
Time Frame: 9 months
Population: 1 participant skipped this measure so overall number is 39 instead of 40
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 39
score on a scale
  Convenience of intervention | 8.79 (1.17)
  Relevance of intervention | 8.46 (1.67)
  Helpfulness of intervention | 8.54 (1.55)

3. Secondary Outcome: PROMIS Satisfaction With Participation in Social Roles - Short Form 8a
Description: Brief measure of satisfaction with ability and participation in activities and roles (e.g., work at home, regular personal and household responsibilities, do things for family) Higher scores indicate more satisfaction with participation. Raw scores range from 8 to 40. 8 items are responded to on a scale of 1 = not at all to 5 = very much.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 40
score on a scale | 21.8 (9.54)

4. Secondary Outcome: Hope - State Hope Scale (Snyder)
Description: Brief measure of agency and pathways thinking. 6 items responded to on a scale of 1 = definitely false to 8 = definitely true. Items are summed for a total score (possible range = 6 - 48). Higher scores indicate higher hope.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 40
total score on a scale | 31.3 (7.9)

5. Secondary Outcome: Purpose - PROMIS Meaning and Purpose 4a
Description: Brief measure assessing one's sense of purpose and that there are reasons for living; 4 items responded to on a scale of 1 = not at all to 5 = very much (possible raw score range = 4 - 20). Higher scores indicate greater meaning and purpose.
Time Frame: 9 months
Population: 1 participant skipped this measure so overall number is 39 instead of 40
Measure: Mean (Standard Deviation); unit: total raw score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 39
total raw score on a scale | 16.4 (3.7)

6. Secondary Outcome: Distress - PROMIS Depression Short Form 6a
Description: Brief measure assessing sense of worthlessness, helplessness, depression, etc. 6 items are responded to on a scale of 1 = never to 5 = always (possible raw scores range from 6-30). Higher scores indicate greater distress.
Time Frame: 9 months
Population: 1 participant skipped this measure so overall number is 39 instead of 40
Measure: Mean (Standard Deviation); unit: total raw score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 39
total raw score on a scale | 11.3 (5.87)

7. Secondary Outcome: Lung Cancer Stigma - Lung Cancer Stigma Inventory (Hamann)
Description: measure of lung cancer stigma. 25 items making up three subscales (perceived stigma, internalized stigma, and constrained disclosure). Items are responded to on a scale of 1 = not at all to 5 = extremely. Items are summed, with a higher score indicating greater lung cancer stigma/worse outcome (possible total score range = 25-125) . Clinical cutoff of a total score of 37.5 is suggested in literature as significant levels of stigma.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Pathways
Number analyzed (Participants) | 40
total score on a scale | 52 (15.7)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Pathways
All-Cause Mortality (participants affected / at risk) | 3/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04161157/Prot_SAP_ICF_000.pdf